CLINICAL TRIAL: NCT01693393
Title: A Phase II Pilot-Study With Low-dose Sandimmun Optoral (Cyclosporin A) for the Treatment of Primary Sjögren Syndrome
Brief Title: Low Dose Cyclosporin A in Primary Sjögren Syndrome
Acronym: CYPRESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Eugen Feist, PD. Dr. med. Eugen Feist, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COLO400BDE02T
Record Dates: First submitted 2012-09-14; First posted 2012-09-26 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Sjögren´s Syndrome
Keywords: primary Sjogren´s Syndrome; Cyclosporine
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclosporine A (Other): All patients will receive Cyclosporine A in a dose of 2mg/kg/BW daily for 16 weeks
  Interventions: Drug: Cyclosporine A

INTERVENTIONS:
Drug: Cyclosporine A — Patients will receive Cyclosporine A in a dose of ca. 2mg/kg/BW daily for a 16 week period
  Other Names: Sandimmun optoral

SUMMARY:
Sandimmun optoral (Cyclosporin A) is used for the musculoskeletal manifestations of Primary Sjögren Syndrome

DETAILED DESCRIPTION:
NSAR are used currently for the treatment of musculoskeletal manifestations at Sjögren Syndrome for the symptomatic release of pain. For therapy-resistant cases drugs also used in Rheumatoid Arthritis are used. For these drugs there is no registration for the treatment of Sjögren Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a primary Sjögren´s Syndrome
* Liver values above 1,5 ULN
* uncontrolled arterial hypertension
* intraarticular or systemic use of Glucocorticoids in the last 4 weeks before
* begin with Study medication

Exclusion Criteria:

* pre-treatment with Cyclosporine A
* Infection
* Neoplasia
* relevant cardiac, pulmonary, neurologic or psychiatric disease
* life-Vaccination within 4 weeks before begin with study medication
* pregnant or breast-feeding
* weight under 45kg or more than 110kg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Examination of the therapeutic effects (improvement in number of tender, swolen joints, DAS 28) of low dose Cyclosporine A in patients with primary Sjögren Syndrome and articular involvement after a treatment-phase of 16 weeks. | 16 weeks

SECONDARY OUTCOMES:
Evaluation of the safety (type and number of adverse events and serious adverse events) of low-dose Cyclosporine A in patients with primary Sjögren Syndrome | 28 weeks

OTHER OUTCOMES:
Study the general health changes and improvement of Sicca-symptoms | 16 weeks
Documentation of improvement of articular manifestations by ultrasound examination | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eugen Feist, Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite Universitätsklinikum Berlin Campus Mitte, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Kedor C, Zernicke J, Hagemann A, Gamboa LM, Callhoff J, Burmester GR, Feist E. A phase II investigator-initiated pilot study with low-dose cyclosporine A for the treatment of articular involvement in primary Sjogren's syndrome. Clin Rheumatol. 2016 Sep;35(9):2203-10. doi: 10.1007/s10067-016-3360-4. Epub 2016 Jul 28. PMID 27470087